CLINICAL TRIAL: NCT01969630
Title: Paclitaxel-eluting Balloon Angioplasty With Provisional Use of Nitinol Stent Versus Systematic Implantation of Paclitaxel-eluting Stent for the Treatment of Femoropopliteal de Novo Lesions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, Director, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Arezzo011
Record Dates: First submitted 2013-10-21; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Peripheral Artery Disease
Keywords: femoropopliteal lesions
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEB (Active Comparator): PEB angioplasty plus provisional nitinol stent implantation
  Interventions: Device: PEB
- PES (Experimental): Systematic PES angioplasty
  Interventions: Device: PES

INTERVENTIONS:
Device: PEB — Paclitaxel eluting balloon angioplasty plus provisional nitinol stent implantation
  Arms: PEB
Device: PES — Systematic Paclitaxel eluting stent angioplasty
  Arms: PES

SUMMARY:
To determine in patients with symptomatic femoropopliteal lesions whether percutaneous revascularization with paclitaxel-eluting balloon angioplasty (PEB) and provisional nitinol stent is superior with respect to the 12-month incidence of restenosis compared to treatment with systematic paclitaxel-eluting stent (PES) angioplasty

ELIGIBILITY:
Inclusion Criteria:

* intermittent claudication or critical limb ischemia
* de novo stenosis ≥ 50% or occlusion of at least 40 mm in length located in femoropopliteal arteries
* presence of a clear healthy segment between the lesion in superficial femoral and common femoral artery and between popliteal and tibioperoneal trunk
* presence of at least 1 patent tibial vessel with distal run-off (below-the-knee artery was considered patent if free from obstructive lesions determining angiographic stenosis >70%)

Exclusion Criteria:

* life expectancy <1 year
* contraindication for combined antiplatelet therapy or known allergy to nickel or paclitaxel
* need for major amputation (MA) at the time of enrolment
* Failure to recanalize intended below-the-knee arteries in CLI patients at risk of major amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
angiographic binary restenosis | 12 months
  incidence of binary restenosis

SECONDARY OUTCOMES:
Composite of all cause mortality, major amputation and target lesion revascularization. | 12 months
  incidence of composite endpoint of all cause mortality, major amputation and target lesion revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy

REFERENCES:
- [Derived] Liistro F, Angioli P, Porto I, Ducci K, Falsini G, Ventoruzzo G, Ricci L, Scatena A, Grotti S, Bolognese L. Drug-Eluting Balloon Versus Drug-Eluting Stent for Complex Femoropopliteal Arterial Lesions: The DRASTICO Study. J Am Coll Cardiol. 2019 Jul 16;74(2):205-215. doi: 10.1016/j.jacc.2019.04.057. PMID 31296293